CLINICAL TRIAL: NCT05042908
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of LBL-003 Injection in Patients With Advanced Malignancies
Brief Title: Evaluation of LBL-003 Phase I Study in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Collaborators: Henan Cancer Hospital (Other Government); Hunan Cancer Hospital (Other); Shandong Cancer Hospital and Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-003-CN-001
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Advanced Malignant Tumor
Keywords: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-003 (Experimental): Drug: LBL-003 injection ; Initial dose - MTD; Q2W
  Interventions: Drug: LBL-003 Injection

INTERVENTIONS:
Drug: LBL-003 Injection — LBL-003 was given every two weeks for treatment
  Other Names: LBL-003

SUMMARY:
This study is a single-arm, dose-escalation phase I clinical trial to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of LBL-003 injection in patients with advanced malignant tumors.

DETAILED DESCRIPTION:
The purpose of the single-dose escalation study of LBL-003 in subjects with advanced malignant tumors was to evaluate the safety and tolerability of monotherapy to determine the MTD (or MAD) and to determine the clinically recommended dose of LBL-003 monotherapy.

All subjects in this study underwent pharmacokinetic (PK) and pharmacodynamic (PD) studies. The dosing frequency of LBL-003 is once every 2 weeks (Q2W), and the subsequent dosing frequency is adjusted according to the obtained PK and tolerability results.

This study is expected to enroll 17-36 patients with solid tumors who have no standard treatment or have treatment failure with standard treatment or are not suitable for standard treatment at this stage.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female aged 18-75 years (including borderline values) at the time of signing the informed consent form;
2. ECOG score: 0-1;
3. Agree to follow the study treatment plan and visit plan, voluntarily enrolls, and signs the written informed consent.
4. Subjects with advanced malignant solid tumors confirmed by histology or cytology have failed the standard treatment or have no standard treatment protocol or are not suitable for standard treatment at this stage.
5. Subjects should have at least one evaluable lesion as defined by RECIST V1.1;
6. Subjects are expected to survive at least 12 weeks;

Exclusion Criteria:

1. History of immunodeficiency, including positive HIV antibody test results；
2. Active hepatitis (hepatitis B or C)；
3. having undergone major surgery or still in the recovery phase of an earlier surgery within 4 weeks before the first administration;
4. Women during pregnancy or lactation;
5. The investigator's assessment that there may be other factors affecting compliance among participants or that some may not be suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Within 4 weeks after receiving the first dose of the test drug
  MTD is defined as the hightest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycles.
Dose-limiting toxicities（DLT） | Within 4 weeks after receiving the first dose of the test drug
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment. It was used to evaluate the safety.

SECONDARY OUTCOMES:
Number of subjcects with adverse events and serious adverse events | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  The safety profile of LBL-003 will be assessed by monitoring the adverse event(AE)
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  Maximum serum concentration
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  After taking a single dose, Time to reach maximum plasma concentration
immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy).
  ORR (including the rates of complete response (CR) and partial response (PR)), evaluated based on the RECIST 1.1, refers to the percentage of study subjects who achieve a complete response or partial response.
Pharmacodynamic (PD) index | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  The evaluation index is receptor occupancy rate in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital
Locations (3):
- China (3):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shangdong Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No